CLINICAL TRIAL: NCT03339999
Title: A Randomized, Double-Blind, Placebo-Controlled, Study to Assess the Efficacy, Safety, Pharmacokinetics and Pharmacodynamics of AGN-242428 in Patients With Plaque Psoriasis
Brief Title: AGN-242428 in the Treatment of Plaque Psoriasis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: safety reason
Sponsor: Vitae Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1957-201-001
Record Dates: First submitted 2017-11-08; First posted 2017-11-13 (Actual); Results first posted 2021-04-06 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-03

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo-matching AGN-242428 capsules, oral administration, once-daily for up to 12 weeks.
  Interventions: Drug: Placebo
- AGN-242428 Higher Dose (Experimental): AGN-242428 capsules, oral administration, once-daily for up to 12 weeks.
  Interventions: Drug: AGN-242428
- AGN-242428 Medium Dose (Experimental): AGN-242428 capsules, oral administration, once-daily for up to 12 weeks.
  Interventions: Drug: AGN-242428
- AGN-242428 Lower Dose (Experimental): AGN-242428 capsule and placebo-matching AGN-242428 capsule, oral administration, once-daily for up to 12 weeks.
  Interventions: Drug: AGN-242428; Drug: Placebo

INTERVENTIONS:
Drug: AGN-242428 — AGN-242428 administered as an oral capsule(s) once daily.
  Arms: AGN-242428 Higher Dose; AGN-242428 Lower Dose; AGN-242428 Medium Dose
Drug: Placebo — Placebo administered as an oral capsule(s) once daily.
  Arms: AGN-242428 Lower Dose; Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, tolerability, pharmacokinetics and pharmacodynamics of 3 doses of AGN-242428 in adult participants with moderate to severe plaque-type psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have a confirmed diagnosis of plaque psoriasis, diagnosed at least 6 months before study with a Physician's Global Assessment (PGA) score ≥ 3 at screening and baseline
* Severity of disease must be at least moderate, defined as Psoriasis Area and Severity Index (PASI) ≥ 12 and % body surface area (BSA) ≥ 10
* Participant is a candidate for phototherapy or systemic therapy for psoriasis
* Body weight of at least 55 kilograms (kg) (121 (pound) lbs)

Exclusion Criteria:

* Non-plaque forms of psoriasis (erythrodermic, guttate, pustular) or drug-induced psoriasis
* Psoriasis which has not been stable for the 4 weeks prior to screening and which is unstable at Study Day 1
* History of Gilbert's, Rotor, or Dubin-Johnson syndromes or any other disorder of bilirubin metabolism
* History of active mycobacterium tuberculosis (TB) infection or untreated or inadequately treated latent TB
* Positive QuantiFERON test for TB infection at screening
* Had a vaccination with Bacillus Calmette-Guérin (BCG) within 12 months prior to baseline
* Positive drug and/or alcohol test at screening (with the exception of marijuana). Retesting in the case of a positive alcohol test is allowed at the discretion of the sponsor
* Current treatment or history of treatment with any anti-Tumor Necrosis Factor alpha (TNFα) biologic therapy within 3 months or 5 half-lives of study, and/or all other biologics within 6 months of study (Day 1)
* Efficacy failure on 2 or more biologic agents for the treatment of psoriasis when the failures occurred within 1 year of the initiation of the therapy of the first biologic agent
* Alanine aminotransferase (ALT), aspartate aminotransferase (AST) or total bilirubin (TBL) exceeding 1.5 times the upper limit of normal (ULN) at screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2018-03-22 (Actual); Study Completion 2018-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christy Harutunian, Study Director — Allergan
Locations (15):
- United States (15):
  - Total Skin and Beauty Dermatology Center, PC, Birmingham, Alabama
  - Radiant Tucson, Tucson, Arizona
  - Johnson Dermatology, Fort Smith, Arkansas
  - First OC Dermatology, Fountain Valley, California
  - University Clinical Trials, San Diego, California
  - Horizons Clinical Research Center, Denver, Colorado
  - Belleair Research Center, Pinellas Park, Florida
  - Dawes Fretzin Dermatology Group, Indianapolis, Indiana
  - The Indiana Clinical Trials Center, PC, Plainfield, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Kansas City Dermatology, Overland Park, Kansas
  - Somerset Skin Centre, Troy, Michigan
  - Oregon Medical Research Center, Portland, Oregon
  - Arlington Research Center, Inc, Arlington, Texas
  - Progressive Clinical Research, San Antonio, Texas

REFERENCES:
- See also: Additional information on study locations near you may be found at AllerganClinicalTrials.com. For any study not on AllerganClinicalTrials.com, please contact IR-CTRegistration@Allergan.com for assistance. — http://AllerganClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: As the study was terminated, no participants completed the planned dosing schedule of 16 weeks.
Period: Overall Study
Arm/Group | Placebo | AGN-242428 Higher Dose | AGN-242428 Medium Dose | AGN-242428 Lower Dose
Started | 7 | 6 | 6 | 5
Modified Intent-to-Treat Population | 7 | 6 | 5 | 4
Safety Population: Received Treatment | 7 | 6 | 6 | 4
Completed | 0 | 0 | 0 | 0
Not Completed | 7 | 6 | 6 | 5
Not completed — Adverse Event | 1 | 2 | 2 | 1
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Study Terminated by Sponsor | 6 | 3 | 4 | 3

BASELINE CHARACTERISTICS:
Population: Modified Intent-to-Treat (mITT) population included all randomized participants with at least 1 postbaseline Psoriasis Area and Severity Index (PASI) assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | AGN-242428 Higher Dose | AGN-242428 Medium Dose | AGN-242428 Lower Dose | Total
Number analyzed (Participants) | 7 | 6 | 5 | 4 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.3 (16.87) | 50.8 (10.83) | 52.0 (10.02) | 44.8 (11.00) | 48.5 (12.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 1 | 0 | 5
  Male | 4 | 5 | 4 | 4 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 5 | 6 | 4 | 4 | 19
  Asian | 2 | 0 | 1 | 0 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 1 | 1 | 7
  Not Hispanic or Latino | 5 | 3 | 4 | 3 | 15
Psoriasis Area and Severity Index (PASI) Score at Baseline [Mean (Standard Deviation); unit: score on a scale] — The PASI score ranges from 0-72 (with a higher score indicating greater severity of psoriasis), based on a combination of the severity (erythema, induration, and desquamation) of psoriasis and percentage of affected area.
  score on a scale | 18.20 (4.819) | 14.37 (3.635) | 18.78 (7.281) | 15.98 (3.699) | 16.88 (5.023)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving a Reduction (Improvement) in Psoriasis Area and Severity Index (PASI) Score of ≥ 75% From Baseline to Week 16
Description: The PASI score ranges from 0-72 (with a higher score indicating greater severity of psoriasis), based on a combination of the severity (erythema, induration, and desquamation) of psoriasis and percentage of affected area.
Time Frame: Baseline (Day 1) to Week 16
Population: No data was collected for this Outcome Measure because the study was terminated and no participants reached the Week 16 timepoint.
Arm/Group | Placebo | AGN-242428 Higher Dose | AGN-242428 Medium Dose | AGN-242428 Lower Dose
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Secondary Outcome: Percentage of Participants Achieving ≥ 2-point Reduction (Improvement) in Physician's Global Assessment (PGA) Score at Week 16
Description: The investigator evaluated the participant's overall severity of psoriasis using the PGA 5-point scale (0 to 4) where 0=Clear and 4=Severe.
Time Frame: Baseline (Day 1) to Week 16
Population: as for outcome 1
Arm/Group | Placebo | AGN-242428 Higher Dose | AGN-242428 Medium Dose | AGN-242428 Lower Dose
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Percentage of Participants Achieving a Clear (0) or Almost Clear (1) Score in PGA at Week 16
Description: The investigator evaluated the participant's overall severity of psoriasis using the PGA 5-point scale (0 to 4) where 0=Clear to 4=Severe.
Time Frame: Week 16
Population: as for outcome 1
Arm/Group | Placebo | AGN-242428 Higher Dose | AGN-242428 Medium Dose | AGN-242428 Lower Dose
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Secondary Outcome: Percentage of Participants Achieving Reduction (Improvement) in PASI Score of ≥ 50% From Baseline to Week 16
Description: as for outcome 1
Time Frame: Baseline (Day 1) to Week 16
Population: as for outcome 1
Arm/Group | Placebo | AGN-242428 Higher Dose | AGN-242428 Medium Dose | AGN-242428 Lower Dose
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Percentage of Participants Achieving Reduction (Improvement) in PASI Score of ≥ 90% From Baseline to Week 16
Description: as for outcome 1
Time Frame: Baseline (Day 1) to Week 16
Population: No data was collected for this Outcome Measure because the study was terminated and no participants reached the Week 16 primary timepoint.
Arm/Group | Placebo | AGN-242428 Higher Dose | AGN-242428 Medium Dose | AGN-242428 Lower Dose
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. An AE was considered a TEAE if the AE began or worsened (increased in severity or became serious) on or after the date of the first dose of study drug.
Time Frame: First dose of study drug to the last dose of study drug (up to Week 12) plus approximately 30 days past last dose
Population: Safety population included all participants who received at least 1 administration of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | AGN-242428 Higher Dose | AGN-242428 Medium Dose | AGN-242428 Lower Dose
Number analyzed (Participants) | 7 | 6 | 6 | 4
Participants | 5 | 3 | 4 | 1

7. Secondary Outcome: Number of Participants With TEAEs Leading to Discontinuation
Description: An AE is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. An AE was considered a TEAE if the AE began or worsened (increased in severity or became serious) on or after the date of the first dose of study drug.
Time Frame: First dose of study drug to the last dose of study drug (up to Week 12) plus approximately 30 days past last dose
Population: Safety population included all participants who received at least 1 administration of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | AGN-242428 Higher Dose | AGN-242428 Medium Dose | AGN-242428 Lower Dose
Number analyzed (Participants) | 7 | 6 | 6 | 4
Participants | 1 | 2 | 2 | 1

8. Secondary Outcome: Number of Participants With TEAEs Considered Related to the Study Treatment as Per Investigator
Description: An AE is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. An AE was considered a TEAE if the AE began or worsened (increased in severity or became serious) on or after the date of the first dose of study drug. The TEAEs related to the study drug, as assessed by Investigator are reported.
Time Frame: First dose of study drug to the last dose of study drug (up to Week 12) plus approximately 30 days past last dose
Population: Safety population included all participants who received at least 1 administration of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | AGN-242428 Higher Dose | AGN-242428 Medium Dose | AGN-242428 Lower Dose
Number analyzed (Participants) | 7 | 6 | 6 | 4
Participants | 1 | 3 | 3 | 1

9. Secondary Outcome: Plasma Concentration of AGN-242428
Time Frame: Single sample predose at Week 4 and 8 Visits, single sample 1-2 hours postdose at Weeks 6 and 10 Visits
Population: Pharmacokinetic (PK) population included all participants who received AGN-242428 and had available plasma concentration data at the given timepoint. No PK data was collected at Week 12 for participants who received AGN-242428 or Week 16 as the study was terminated.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | AGN-242428 Higher Dose | AGN-242428 Medium Dose | AGN-242428 Lower Dose
Number analyzed (Participants) | 5 | 4 | 3
ng/mL
  Week 4: number analyzed (Participants) | 5 | 3 | 3
  Week 4 | 1500 (692) | 1060 (449) | 488 (125)
  Week 6: number analyzed (Participants) | 1 | 4 | 2
  Week 6 | 3720 (NA) — Standard deviation was not calculated due to limited PK data. | 1150 (881) | 718 (NA) — Standard deviation was not calculated due to limited PK data.
  Week 8: number analyzed (Participants) | 1 | 3 | 2
  Week 8 | 1300 (NA) — Standard deviation was not calculated due to limited PK data. | 886 (376) | 616 (NA) — Standard deviation was not calculated due to limited PK data.
  Week 10: number analyzed (Participants) | 0 | 1 | 0
  Week 10 |  | 483 (NA) — Standard deviation was not calculated due to limited PK data. |
  Week 12: number analyzed (Participants) | 0 | 0 | 0
  Week 16: number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: First dose of study drug to the last dose of study drug (up to Week 12) plus approximately 30 days past last dose
Description: Safety population included all participants who received at least 1 administration of study treatment.
Arm/Group | Placebo | AGN-242428 Higher Dose | AGN-242428 Medium Dose | AGN-242428 Lower Dose
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/6 | 0/6 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6 | 0/6 | 0/4
Other Adverse Events (participants affected / at risk) | 5/7 | 3/6 | 4/6 | 1/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=7) | AGN-242428 Higher Dose (N=6) | AGN-242428 Medium Dose (N=6) | AGN-242428 Lower Dose (N=4)
Nausea (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 2 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 0 | 1
Mycobacterium tuberculosis complex test positive (Investigations) | 0 | 0 | 1 | 0
Transaminases increased (Investigations) | 0 | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 2 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Glycosuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2017-12-21): https://cdn.clinicaltrials.gov/large-docs/99/NCT03339999/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-16): https://cdn.clinicaltrials.gov/large-docs/99/NCT03339999/SAP_001.pdf